CLINICAL TRIAL: NCT02750098
Title: Comparison of Aqueous and Plasma Glucose Level in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Irina Barequet, Cornea and refractive surgery specialist, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 296416
Record Dates: First submitted 2016-04-11; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus, Cataract, Aqueous humor
MeSH Terms: conditions — Diabetes Mellitus; Cataract

ARMS (1):
- Diabetic patients (Experimental): Diabetic patients planned to undergo elective cataract surgery
  Interventions: Other: Glucose measurement

INTERVENTIONS:
Other: Glucose measurement — 1. Elective cataract surgery
  2. Blood glucose measurement - glucometer
  3. Aqueous humor glucose measurement - at beginning of cataract surgery - glucometer
  4. Perioperative Hemoglobin A1c level - blood laboratory test

SUMMARY:
Comparison of aqueous and plasma glucose level in diabetic patients

High glucose concentrations in aqueous humor are thought to be related of diabetic ocular injury, including cataract and diabetic keratopathy. The primary mechanisms are nonenzymatic glycation, oxidative stress and activation of polyol pathway. However, glucose concentrations in aqueous humor of diabetic patients was only examined in a few patients in the past.

This study will compare glucose concentration in blood plasma and aqueous humor in diabetic patients undergoing cataract surgery. Perioperative Hemoglobin A1c concentrations will also be examined. Correlation between these parameters will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

- Diabetic patients planed for elective cataract surgery

Exclusion Criteria:

* s/p traumatic eye injury
* past or current uveitis
* patients using prescription eye drops except lubricants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Aqueous humor glucose concentration | Day of cataract surgery

SECONDARY OUTCOMES:
Plasma glucose concentrations | Day of cataract surgery
Hemoglobin A1c | Perioperative month